CLINICAL TRIAL: NCT07048262
Title: A Phase 2b, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose Range Finding Study to Evaluate the Efficacy, Safety, and Tolerability of Nebulized CSL787 in Adults (18 to 85 Years) With Non-cystic Fibrosis Bronchiectasis
Brief Title: Dose Range Finding, Efficacy, and Safety Study of Nebulized CSL787 in Adults With Non-cystic Fibrosis Bronchiectasis (NCFB)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL787_2001; 2024-518821-13-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: Chronic respiratory disease; Inflammation; Chronic bacterial infection
MeSH Terms: conditions — Inflammation | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, parallel-group, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- CSL787 High Dose (Experimental): Participants in this arm will receive a high dose of CSL787.
  Interventions: Biological: CSL787; Device: Nebulizer
- CSL787 Low Dose (Experimental): Participants in this arm will receive a low dose of CSL787.
  Interventions: Biological: CSL787; Device: Nebulizer
- Placebo (Placebo Comparator): Participants in this arm will receive placebo.
  Interventions: Drug: Placebo; Device: Nebulizer

INTERVENTIONS:
Biological: CSL787 — CSL787 high or low doses once daily (QD) will be administered via inhalation over a period of 6 to 12 months.
  Arms: CSL787 High Dose; CSL787 Low Dose
Drug: Placebo — Participants will receive a matching volume of placebo QD over a period of 6 to 12 months.
  Arms: Placebo
Device: Nebulizer — The nebulizer is a CE-marked device.

SUMMARY:
This study is a phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose range finding study designed to explore the efficacy, safety, and tolerability of 2 active treatment regimens of CSL787 (immunoglobulin G [IgG] inhalation solution) compared with placebo over a period of 6 to 12 months independent of the occurrence of pulmonary exacerbations.

The primary aim of the study is to characterize the overall effect of CSL787 as well as the dose response of 2 active treatment regimens of inhaled CSL787 administered to participants with NCFB toward prolonging the TTF exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Adult between the ages of 18 to 85 years
* Primary diagnosis of NCFB confirmed by chest computed tomography (CT) scan, where bronchiectasis has been documented by a radiologist. Diagnosis in the medical records based on historical scans is acceptable if the chest CT scan confirming the participant's NCFB diagnosis was performed within 12 months before enrollment. Participants for whom no chest CT scan results are available within the previous 12 months will undergo a chest CT scan during the Screening Period
* Exacerbation history within the previous 1 year defined as either 1 of the following:
* >= 2 documented exacerbations requiring oral and/or intravenous (IV) antibiotic therapy to treat a pulmonary infection.

OR

* 1 documented exacerbation requiring oral and/or IV antibiotic therapy to treat a pulmonary infection and a St. George's Respiratory Questionnaire (SGRQ) Symptoms score of > 40 at Screening.
* Note: Other medications to treat NCFB such as: oral macrolides, or dipeptidyl peptidase-1 (DPP-1) inhibitors are allowed, provided >= 1 historical exacerbation occurred while on the medication for >= 3 months at a stable dose.
* Postbronchodilator percentage of the predicted normal forced expiratory volume in 1 second of expiration [FEV1% predicted] > 35% and forced expiratory volume in 1 second (FEV1) >= 1 liter (L) obtained in accordance with American Thoracic Society (ATS) / European Respiratory Society (ERS) standards for spirometry during Screening and at Baseline.

Exclusion Criteria:

* History of bronchospasm in response to inhaled therapies including inhaled antibiotics
* Known or suspected hypersensitivity, or other severe reactions, to the investigational product (IP), to any excipients of the IP, or to other immunoglobulin.
* Primary diagnosis of other pulmonary disorders, including chronic obstructive pulmonary disease (COPD) asthma or, diffuse panbronchiolitis (DPB), as determined by the investigator.
* Pulmonary exacerbation requiring antibiotic therapy within the 4 weeks before Baseline.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Time to first (TTF) Exacerbation | Up to Month 12
  TTF exacerbation, where an exacerbation is defined as a deterioration in >= 3 of the following symptoms for >= 48 hours: cough; sputum volume and / or consistency; sputum purulence; breathlessness and / or exercise tolerance; fatigue and / or malaise; hemoptysis AND a clinician determines that antibiotic therapy is required.

SECONDARY OUTCOMES:
Annualized Exacerbation Rate (AER) (Exacerbation Event Rate Per-participant Year) | Up to Month 12
Number of Participants Achieving a Clinically Important Difference in the Quality of Life-Bronchiectasis (QoL-B) Respiratory Symptoms Scale | Up to Month 12
  The QoL-B questionnaire is a self-administered measure assessing symptoms, functioning, and health-related quality of life for patients with NCFB. This questionnaire contains 37 items on 8 different scales (Respiratory symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions, and Treatment Burden). For each scale, scores are standardized on a 0-to-100-point scale; higher scores indicate better health-related quality of life.
Percentage of Participants Achieving a Clinically Important Difference in the QoL-B Respiratory Symptoms Scale | Up to Month 12
  The QoL-B questionnaire is a self-administered measure assessing symptoms, functioning, and health-related quality of life for patients with NCFB. This questionnaire contains 37 items on 8 different scales (Respiratory symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions, and Treatment Burden). For each scale, scores are standardized on a 0-to-100-point scale; higher scores indicate better health-related quality of life.
Change From Baseline in QoL-B Respiratory Symptoms Scale | From Baseline to Months 6 and 12
  The QoL-B questionnaire is a self-administered measure assessing symptoms, functioning, and health-related quality of life for patients with NCFB. This questionnaire contains 37 items on 8 different scales (Respiratory symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions, and Treatment Burden). For each scale, scores are standardized on a 0-to-100-point scale; higher scores indicate better health-related quality of life.
Change From Baseline in Total Colony-forming Unit (CFUs) for Pathogenic Bacteria Isolated from Sputum | From Baseline to Month 1
Number of Participants with Treatment-emergent Adverse events (TEAEs) and Serious Adverse Events (SAEs) | Up to Month 13
Percentage of Participants with TEAEs and SAEs | Up to Month 13

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (13):
- Australia (2):
  - The Prince Charles Hospital, Queensland
  - Westmead Hospital, Westmead
- Japan (11):
  - Fukuoka University Chikushi Hopsital, Chikushino-shi
  - Kyusho Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka
  - Ibaraki Prefectural Central Hospital, Ibaraki
  - Kazunori Tobino Iizuka Hospital, Iizuka-shi
  - National Hospital Organization Minami Kyoto Hospital, Kyoto
  - Matsusaka Municipal Hospital, Mie
  - National Hospital Organization Kinki Chuo Chest Medical Center, Osaka
  - Shimonoseki City Hospital, Shimonoseki-shi
  - Japan Anti-Tuberculosis Association, Fukujuji Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - National Hospital Organization Mie Chuo Medical Center, Tsu

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e. FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.